CLINICAL TRIAL: NCT07322341
Title: A Phase 2 Trial of SX-682 and Atezolizumab in Patients With Advanced NSCLC Who Progressed on Prior Chemotherapy and Immune Checkpoint Inhibitor (ICI) Therapy
Brief Title: SX-682 and Atezolizumab for the Treatment of Advanced or Metastatic, Recurrent Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Genentech, Inc. (Industry); Syntrix Biosystems, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1125839; NCI-2025-09043 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P50CA228944-07A1 (NIH)
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Specimen Handling; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SX-682 and atezolizumab) (Experimental): Patients receive SX-682 PO BID on days -7 - 21 of cycle 1 and on days 1-21 of each cycle thereafter and atezolizumab SC on day 1 of each cycle. Cycles repeat every 21 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients undergo brain MRI during screening and CT scan or MRI, blood sample collection and tumor biopsy on trial and may undergo at screening.
  Interventions: Biological: Atezolizumab; Drug: CXCR1/2 Inhibitor SX-682; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biopsy Procedure

INTERVENTIONS:
Biological: Atezolizumab — Given SC
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Drug: CXCR1/2 Inhibitor SX-682 — Given PO
  Other Names: SX 682; SX-682; SX682
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Bx

SUMMARY:
This phase II trial tests how well SX-682 and atezolizumab works for the treatment of non-small cell lung cancer (NSCLC) that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic), and has come back after a period of improvement (recurrent). SX-682 blocks proteins that may be able to stimulate the immune system to kill and eliminate tumor cells. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving SX-682 and atezolizumab may be effective for the treatment of advanced or metastatic, recurrent NSCLC.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive SX-682 orally (PO) twice daily (BID) on days -7 - 21 of cycle 1 and on days 1-21 of each cycle thereafter and atezolizumab subcutaneously (SC) on day 1 of each cycle. Cycles repeat every 21 days for up to 5 years in the absence of disease progression or unacceptable toxicity. Patients undergo brain magnetic resonance imaging (MRI) during screening and computed tomography (CT) scan or MRI, blood sample collection and tumor biopsy on trial and may undergo at screening.

After completion of study treatment, patients are followed up within 30 days if treatment is discontinued for safety, disease progression, or early withdrawal and every 12 weeks for up to 84 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Ability to understand and willingness to sign a written informed consent document
* Pathologically or cytologically confirmed non-small cell lung cancer with no known oncogenic EGFR mutation, ALK fusion, ROS1 fusion or RET fusions.

  * For participants with NSCLC harboring an oncogenic alteration other than the above must have received prior targeted therapy (e.g. small molecule inhibitor therapy or antibody drug conjugates). A wash-out of at least 5 half-lives is required prior to start of study treatment
* Metastatic or recurrent NSCLC. Stage 3C per 8th edition TNM stage classification is allowed if not amenable to curative surgery or radiation per investigator judgment
* Participants must have received and progressed on at least 6 weeks of treatment with prior anti-PD-1 or anti-PD-L1 therapy for advanced disease. Also, participants must have received prior platinum doublet chemotherapy. Anti-PD1/PD-L1 therapy may have been received concurrently with chemotherapy or as sequential therapy (e.g. anti-PD1 followed by chemotherapy).

  * For participants who received neoadjuvant, adjuvant and/or consolidation anti-PD-1 or anti-PD-L1 therapy for stage 1 - 3 NSCLC: If they experienced disease progression ≤ 365 days from initiation of anti-PD-1 or anti-PD-L1 therapy, this counts as the allowed anti-PD-1 or anti-PD-L1 therapy for advanced disease.
  * For participants who experienced disease progression more than 365 days from initiation of anti-PD-1 or anti-PD-L1 therapy for advanced disease, this is not considered anti-PD-1 or anti-PD-L1 therapy for advanced disease. These patients must have received anti-PD-1 or anti-PD-L1 therapy for stage 4 or recurrent disease
* Participants must have a minimum of 28 days after the last dose, or 5 half-lives of washout period (whichever is shorter) from last dose of most recent systemic therapy prior to initiation of study treatment, including investigational agents
* Participants must have at least one site of measurable disease as determined by the investigator, using RECIST v 1.1 criteria documented within 28 days prior to study treatment initiation
* Participants must have Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1 at the time of informed consent and at the time of treatment initiation
* Participants must be willing to provide pre-treatment archived specimen (taken within a year of trial entry) or undergo a biopsy procedure if archived specimen is not available.

  * If biopsy is not deemed safe, it may be waived after discussion with principal investigator (PI)
* Participants must be willing to provide an on-treatment biopsy, to be obtained at 6 - 9 weeks, if deemed safe by the treating physician
* Platelet count > 100,000/μL
* Absolute neutrophil count > 1,500/μL
* Hemoglobin > 9.0 g/dL. Participants may be transfused to meet this criterion
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) < 2.5 times upper limit of normal
* Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) with the following exception: Patients with known Gilbert disease: serum bilirubin ≥ 3 x ULN
* Creatinine clearance ≥ 30 mL/min
* For patients not receiving therapeutic anticoagulation: International normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Participants of child-bearing potential and sexually active men must agree to use adequate contraception (hormonal methods must be supplemented by barrier method) prior to treatment initiation, during treatment, and for 5 months after the last dose of atezolizumab
* Negative beta human chorionic gonadotropin (β-hCG) pregnancy test result within 14 days prior to initiation of study treatment for participants of childbearing potential. Pregnant or breast-feeding women or intention of becoming pregnant during study treatment or within 5 months of last dose of atezolizumab are not eligible

Exclusion Criteria:

* Presence of other active cancers within the last 2 years. Participants with another cancer who have received definitive therapy at least 2 years previously and no evidence of recurrence are eligible. All participants with previously treated in situ carcinoma are eligible, as are participants with history of non-melanoma skin cancer
* Symptomatic central nervous system (CNS) metastases; participants with known brain metastasis must be asymptomatic with no ongoing requirement for steroids within 7 days prior to start of study treatment, no history of intracranial hemorrhage or spinal cord hemorrhage. If the patient is receiving anti-convulsant therapy, the dose is considered stable

  * Participants with untreated CNS metastases may be enrolled as long as they meet the above criteria. Participants with bulky CNS metastases should consider receiving radiation prior to study entry per investigator judgment
* Participants with spinal cord compression must have received local treatment and must have been symptomatically stable with no use of steroids for at least 7 days prior to start of study treatment
* Participants must not have an active autoimmune disease that has required immune modulating treatment within 1 year prior to consenting (i.e., disease modifying agents, long term corticosteroids). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed. Short-term steroid therapy (≤ 2 weeks) is allowed
* Inability to discontinue corticosteroid therapy; steroids must be tapered off 7 days prior to first dose of SX-682. Limited steroid use for allergic reactions is acceptable
* Known history of primary immunodeficiency
* History of organ transplant or prior allogenic stem cell transplantation that requires use of immunosuppressives
* Current symptomatic pneumonitis and any past history of immune checkpoint inhibitor related pneumonitis regardless of steroid treatment history
* Prior history of grade 3 or higher immune checkpoint inhibitor (ICI)-induced immune-related adverse event (AE) (immune related adverse event [irAE]) except endocrine irAEs that are resolved or managed with replacement therapy
* Radiotherapy within 7 days of start of study treatment
* Major surgery within 21 days of start of study treatment. Minor surgery within 2 weeks of start of study treatment.

  * Placement of vascular access device and biopsies are not considered major or minor surgery and are allowed
* Electrocardiogram (ECG) demonstrating a Fridericia's corrected QT interval (QTcF) interval > 480 msec or patients with congenital long QT syndrome
* Severe lung disease (e.g. chronic obstructive pulmonary disease [COPD]) who cannot stop steroids 7 days prior to start of study treatment
* Serious cerebrovascular and cardiac disease defined as:

  * Active unstable angina pectoris
  * Congestive heart failure New York Heart Association (NYHA) > grade 3
  * Acute myocardial infarction within 3 months of consenting
  * Stroke or transient ischemic attack within 3 months of consenting
* Known active chronic infections: Active hepatitis B, hepatitis C and tuberculosis. Testing is not required for assessment of eligibility per investigator judgment. Active infection requiring IV antibiotics within 7 days of study treatment initiation.

  * Hepatitis C virus (HCV) infection: Patients with known history of HCV infection are eligible if HCV viral load is below the limit of quantification per local assay per investigator judgment.
  * Hepatitis B virus (HBV) infection: Patients with known history of HBV infection are eligible if HBV viral load is below the limit of quantification and negative hepatitis B surface antigen (HBsAg) per local assay per investigator judgment
* Known uncontrolled HIV (human immunodeficiency virus) infection

  * Participants with known HIV infection are allowed if they are receiving anti-retroviral therapy, have CD4+ T-cell count > 350 cells/µL within 6 months prior to study treatment initiation and no history of AIDS- defining opportunistic infection
* Any serious or uncontrolled concomitant disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
* History of leptomeningeal disease
* Treatment with investigational therapy within 28 days prior to initiation of study treatment, or 5 half-lives of washout period (whichever is shorter) from last dose of most recent systemic therapy
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Known allergy or hypersensitivity to any component of the atezolizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2030-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 5 years from treatment initiation
  Response by Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST).

SECONDARY OUTCOMES:
Response rate in the subset of participants with circulating IL-8 levels greater than or equal to 23 pg/ml | Up to 5 years from treatment initiation
  Response by iRECIST. Will be summarized along with 80% confidence intervals.
Duration of response | From date of first documentation of response to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause among participants who achieve a up to 7 years from treatment initiation
  Will be estimated using the method of Kaplan-Meier.
Disease control rate | At 16 weeks
  Defined as immune mediated complete response, immune mediated partial response, confirmed and unconfirmed, immune mediated stable disease.
Response by Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 5 years from treatment initiation
  Defined as complete response and partial response (confirmed and unconfirmed), stable disease.
Progression free survival | From date of start of protocol treatment to date of first documentation of progression, assessed by local review or symptomatic deterioration or death due to any cause, up to 5 years from treatment initiation
  Will be estimated using the method of Kaplan-Meier.
Overall survival | From date of start of protocol treatment to date of death due to any cause, up to 7 years from treatment initiation
  Will be estimated using the method of Kaplan-Meier.
Incidence of adverse events | Up to 5 years from treatment initiation
  As measured by Common Terminology Criteria for Adverse Events version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Baik, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No